CLINICAL TRIAL: NCT02259101
Title: A Randomized Controlled Trial of Cognitive Behavior Therapy for Insomnia With Persons Living With HIV/AIDS
Brief Title: RCT of CBT for Insomnia With PLWHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amit Shahane, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00065796
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Insomnia; HIV; Aids
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I Treatment Condition (Experimental): The CBT-I treatment condition will be delivered in a one-hour per week group format (10 participants) occurring over the course of six-weeks. Four total CBT-I groups occurring over the course of two years will be implemented, with at total of 40 participants enrolled for the CBT-I condition.
  Interventions: Behavioral: CBT-I Treatment Condition
- SH Comparison Condition (Active Comparator): The SH comparison condition will also be delivered in a one-hour per week group format (10 participants) occurring over the course of six-weeks. Four total SH groups over the course of two years will be conducted, with a total of 40 participants enrolled for the SH condition.
  Interventions: Behavioral: SH Comparison Condition

INTERVENTIONS:
Behavioral: CBT-I Treatment Condition — Each group will last approximately 1 hour and will involve completing surveys in order to track both the quantity and quality of sleep. Blood will be drawn twice in order to compare how the body responds to medical illnesses.
  Arms: CBT-I Treatment Condition
Behavioral: SH Comparison Condition — Each group will last approximately 1 hour and will involve completing surveys in order to track both the quantity and quality of sleep. Blood will be drawn twice in order to compare how the body responds to medical illnesses.
  Arms: SH Comparison Condition

SUMMARY:
The proposed study will consist of a randomized controlled trial (RCT) comparing a known efficacious treatment for insomnia (CBT-I) to a sleep hygiene (SH) comparison condition.

DETAILED DESCRIPTION:
The purpose of this study is to test whether a group cognitive-behavioral treatment program for insomnia (CBT-I) will help adults diagnosed with HIV to improve the quantity (number of hours) and the quality of their sleep. The PI will compare adults who participated in the CBT-I program to adults who participated in a Sleep Hygiene group, a common treatment for insomnia. The PI will look at the overall quality of life, and number of hours and quality of sleep of adults who participated in the CBT-I program versus adults in the Sleep Hygiene group. Also, the PI will draw blood to compare how the body responds to medical illnesses between adults in the CBT-I program to adults in the Sleep Hygiene group.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking individuals
* over the age of 18 years old with a diagnosis of HIV or AIDS who is receiving medical care at the Grady Health System's Infectious Disease Program (IDP)
* study subjects must meet the criteria for primary or secondary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision
* must experience difficulty initiating or maintaining non-restorative sleep for at least l month (DSM- IV-TR)
* the sleep disturbance causes clinically significant impairment or distress in important areas of functioning
* sleep efficiency of less than 85%, sleep disturbances that occur three or more days per week, and sleep latency (i.e., time awake after sleep onset greater than 30 minutes)

Exclusion Criteria:

* current substance dependence (within the past six months)
* active psychosis
* Bipolar I and II disorders
* neurocognitive impairment and/or a current diagnosis of dementia
* lack of independent housing
* previous participation in a CBT-I program
* employment in a job requiring shift work that impairs the ability to establish a regular sleep schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Insomnia Symptoms | baseline, up to 5 weeks post-intervention
  Compare insomnia scores on the Insomnia Severity Index (questionnaire) between the CBT-I treatment condition vs. SH comparison condition.

SECONDARY OUTCOMES:
Quality of Life | baseline, up to 5 weeks post-intervention
  Compare quality of life scores on the HIV/AIDS Targeted-Quality of Life (scale) between CBT-I treatment condition vs. SH comparison condition.
Blood Sample | baseline, up to 5 weeks post-intervention
  Evaluate and compare markers of inflammation between participants in the CBT-I treatment condition vs. SH comparison condition.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Shahane, Ph.D., Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital/Infectious Disease Program, Atlanta, Georgia, United States